CLINICAL TRIAL: NCT01917565
Title: The Use of Airtraq Laryngoscope Versus Macintosh Laryngoscope and Fiberoptic Bronchoscope by Experienced Anesthesiologists
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Marmara University (Other)
Responsible Party: Principal Investigator, tolga saracoglu, Assist. Prof. Dr., Marmara University
Other Study IDs: 09.2011.0127
Record Dates: First submitted 2013-08-02; First posted 2013-08-06 (Estimated); Last update posted 2013-08-06 (Estimated); Status verified 2013-08

CONDITIONS: the Hemodynamic Parameters; Intubation Times; Complications During and After Intubation
Keywords: airway management; laryngoscope; Airtraq; Macintosh laryngoscope; fiberoptic bronchoscope; intubation

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional

GROUPS / COHORTS (3):
- Airtraq laryngoscope group: The patients who will be intubated by using Airtraq laryngoscope
- Macintosh laryngoscope group: The patients who will be intubated by using Macintosh laryngoscope
- Fiberoptic bronchoscope group: The patients who will be intubated by using Fiberoptic bronchoscope

SUMMARY:
The investigators hypothesize that when used by experienced anesthesiologists, Airtraq laryngoscope will increase the first-attempt success rate with shorter intubation times and more stable hemodynamic parameters.

DETAILED DESCRIPTION:
The special design of the Airtraq allows the direct exposure of the glottic opening without the necessity of optimal alignment of the oral, pharyngeal and laryngeal axes. The results of the meta-analysis comparing the Airtraq with the conventional Macintosh laryngoscope concluded that the use of Airtraq results in a rapid and accurate intubation. The main advantages of the fiberoptic bronchoscope are minimal airway trauma and minimal deterioration of the hemodynamic parameters.

The purpose of this study is to compare the hemodynamic parameters, intubation times, complications during and after intubation and postoperative sore throat scores of the patients having normal airway anatomy, intubated with Airtraq, Macintosh laryngoscope or fiberoptic bronchoscope, by experienced anesthesiologists.

ELIGIBILITY:
Inclusion Criteria:

* ASA physical status classification of 1 or 2, undergoing elective surgery under general anesthesia and requiring endotracheal intubation

Exclusion Criteria:

* Patients with ASA 3 or 4, Mallampati score of 3 or 4, history of difficult intubation, thyromental distance less than 6.5 cm, sternomental distance less than 12.5 cm, body mass index higher than 35 kg/m2 and limited neck mobility

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients undergoing surgery under general anesthesia
Sampling Method: Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2013-08; Primary Completion 2014-02 (Estimated); Study Completion 2014-03 (Estimated)

PRIMARY OUTCOMES:
The required time to successful tracheal intubation | six months
  The primary outcome variable is the required time to successful tracheal intubation

SECONDARY OUTCOMES:
The first-attempt success rate of tracheal intubation | six months
  The secondary outcome variable is the first-attempt success rate of tracheal intubation

OTHER OUTCOMES:
the effects of the tracheal intubation on hemodynamic parameters | six months
  The other outcome variable is the effects of the tracheal intubation on hemodynamic parameters

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesiology, Marmara University School of Medicine, Istanbul, Turkey (Türkiye)